CLINICAL TRIAL: NCT00003388
Title: A Phase II Study of Doxil (Liposomal Doxorubicin), Cyclophosphamide, Vincristine and Prednisone for AIDS-Related Systemic Lymphoma
Brief Title: Combination Chemotherapy in Treating Patients With AIDS-Related Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Group Chair, Eastern Cooperative Oncology Group
Purpose: Treatment
Other Study IDs: CDR0000066385; E-3D97
Record Dates: First submitted 1999-11-01; First posted 2003-12-02 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Lymphoma
Keywords: AIDS-related peripheral/systemic lymphoma; AIDS-related diffuse large cell lymphoma; AIDS-related immunoblastic large cell lymphoma; AIDS-related small noncleaved cell lymphoma; AIDS-related diffuse mixed cell lymphoma; AIDS-related diffuse small cleaved cell lymphoma; AIDS-related lymphoblastic lymphoma; anaplastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large-Cell, Anaplastic | interventions — Filgrastim; Cyclophosphamide; Cytarabine; Methotrexate; Prednisone; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: filgrastim
Drug: cyclophosphamide
Drug: cytarabine
Drug: methotrexate
Drug: pegylated liposomal doxorubicin hydrochloride
Drug: prednisone
Drug: vincristine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy consisting of liposomal doxorubicin, cyclophosphamide, vincristine, and prednisone in treating patients with AIDS-related lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the one year survival and complete response rate of patients treated with doxorubicin HCl liposome/cyclophosphamide/vincristine/prednisone (Doxil-CVP) for AIDS-related lymphoma. II. Evaluate the toxicity of a combination chemotherapy regimen, Doxil-CVP, in this patient population. III. Evaluate the progression free and overall survival after treatment with Doxil-CVP in this patient population. IV. Evaluate the effects of treatment with Doxil-CVP on plasma viral mRNA levels, CD4+ lymphocyte count, and the incidences and types of opportunistic infections in this patient population.

OUTLINE: Patients are stratified according to disease characteristics. All patients receive a 30 minute infusion of doxorubicin HCl liposome IV, cyclophosphamide IV, and vincristine IV on day 1. Patients also receive oral prednisone on days 1-5. Filgrastim (G-CSF) is administered subcutaneously starting on day 6 and continues until the absolute neutrophil count is at least 10,000/mm3. Treatment courses are repeated every 21 days. Patients with lymphomatous bone marrow involvement and/or category J lymphoma receive cytarabine and methotrexate intrathecally weekly for 4 weeks. Patients with lymphomatous meningitis receive whole brain irradiation and an alternating intrathecal chemotherapy regimen. A minimum of 4 and a maximum of 8 courses are administered. Patients are removed from the study for progressive disease, stable disease after 4 courses, a life threatening infection that would delay treatment for more than 6 weeks, or any delay, except due to neutropenia, in chemotherapy treatment for more than 6 weeks. Patients who achieve a complete response receive an additional 2 courses of therapy. Patients are followed every 3 months for 2 years, every 6 months for 3 years, and annually thereafter.

PROJECTED ACCRUAL: A total of 38 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed AIDS-related non-Hodgkin's lymphoma of the intermediate or high grade histologic types Anaplastic large cell lymphoma allowed Must be HIV positive Must have at least one objective measurable or evaluable disease parameter No parenchymal CNS involvement by lymphoma (meningeal lymphoma allowed) A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: (Except patients with lymphomatous marrow involvement) Absolute neutrophil count at least 1000/mm3 Platelet count at least 50,000/mm3 Hepatic: Bilirubin no greater than 5.0 mg/dL Renal: Creatinine less than 3.0 mg/dL Cardiovascular: Patients with history of heart disease, evidence of congestive heart failure, radiographic evidence of cardiomegaly, or electrocardiographic evidence of a prior myocardial infarction must have LVEF at least at lower limit of normal Neurologic: No grade 3 or greater peripheral neuropathy Other: No prior or concurrent malignancy other than Kaposi's sarcoma, curatively treated basal cell or squamous cell carcinoma of the skin, or curatively treated carcinoma in situ of the cervix Not pregnant or nursing Fertile patients must use effective contraception No history of sensitivity to E. coli-derived proteins

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 5 days since interferon therapy Chemotherapy: No prior cytotoxic chemotherapy except for mucocutaneous Kaposi's sarcoma At least 12 months since cytotoxic chemotherapy for Kaposi's sarcoma Endocrine therapy: Prior steroids allowed No concurrent steroid therapy greater than 5 mg prednisone (or equivalent) per day Radiotherapy: No prior radiotherapy except for mucocutaneous Kaposi's sarcoma Surgery: Not specified Other: No concurrent zidovudine (AZT) Concurrent antiretroviral medications other than AZT allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 1999-07-26 (Actual); Primary Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D. Volm, MD, Study Chair — NYU Langone Health
Locations (5):
- United States (5):
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - Raritan Bay Medical Center, Perth Amboy, New Jersey
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - MBCCOP-Our Lady of Mercy Cancer Center, The Bronx, New York